CLINICAL TRIAL: NCT05482581
Title: The Impact of Policies Regarding E-cigarette(Trial) on Adolescents and Young Adults' Cognition and Behavior for E-cigarette: A Convergent Parallel Mixed-method Study Based on KABP Model.
Brief Title: The Impact of Policies Regarding E-cigarette on Adolescents and Young Adults' Cognition and Behavior for E-cigarette
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Wei XIA, PhD, Associate Professor, Sun Yat-sen University
Other Study IDs: wjn-ChiCTR2200060895
Record Dates: First submitted 2022-07-24; First posted 2022-08-01 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2023-02

CONDITIONS: E-Cig Use
Keywords: Adolescent; Young adult; Policy; Surveys and questionnaires; Qualitative study; Electronic Nicotine Delivery Systems; KABP model; Network epidemiology
MeSH Terms: conditions — Vaping

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Questionnaires assessed adolescents and young adults: ①14-35 years old; ②Being able to read and communicate in Chinese.
  Interventions: Other: Questionnaires set

INTERVENTIONS:
Other: Questionnaires set — Participants will be asked to respond to the demographic information sheet,e-cigarette using characteristics sheet,awareness of e-cigarettes sheet;,willingness to use e-cigarettes sheet, knowledge, attitudes and cognitions related to e-cigarettes sheet, awareness of new regulations on e-cigarette control sheet.

SUMMARY:
Based on the Knowledge，Attitude，Belief and Practice model(KABP model), this study intends to use a mixed method to explore the influencing mechanism of youth and adolescents' cognition and behavior for e-cigarette before and after the promulgation of the new regulations on e-cigarette . Information from network epidemiology (including network links, text, images, audio, video, etc.) was captured to expand the data abundance, and the retrieval behavior of e-cigarettes and the trajectory changes of e-cigarette-related events were explored. Finally, summarize the data, integrate and explain the influencing mechanism of youth and adolescents' attention and cognition on e-cigarette, and provide ideas for subsequent e-cigarette control, as well as theoretical and practical basis for relevant departments to formulate corresponding policies.

DETAILED DESCRIPTION:
Mixed method will be used: the cross-sectional surveys will be conducted on the demographic characteristics, e-cigarette use intentions, e-cigarette use behaviors, attitudes towards e-cigarette , knowledge of e-cigarette harm, reasons for using e-cigarette and the degree of understanding of the new regulations on e-cigarette control ; semi-structured interviews will be conducted with some young people and adolescents interviewed by using phenomenology and qualitative research methods, and the content of the interview will be summarized and analyzed. The primary and secondary categories and dimensions are coded; the analysis results of quantitative data and qualitative data are combined to explain the influencing mechanism of the trial implementation of e-cigarette regulatory regulations on youth and adolescents' cognition of electronic cigarettes and changes in their use behaviors.

Using the network epidemiological method, use the "drop-down word deep mining function" of the 5188 marketing big data website to obtain the relevant keywords of "electronic cigarette", and use the Baidu index and 360 index tools to explore the retrieval behavior of electronic cigarettes and related electronic cigarettes Event trace changes.

Combined with online epidemiological data and mixed method study results, summarize the changes in youth and adolescents' cognition and use of e-cigarettes before and after the promulgation of the new regulations, and provide a theoretical basis for formulating e-cigarette control policies in the future.

ELIGIBILITY:
Inclusion Criteria:

* 14-35 years old;
* Being able to read and write in Chinese.

Exclusion Criteria:

* Those who are unable to communicate due to serious mental or physical illnesses such as deafness, unclear consciousness due to mental illness, etc.

Ages: 14 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Using an online and offline multi-channel model, participants who meet the eligibility criteria are invited to join the study.
Sampling Method: Non-Probability Sample
Enrollment: 453 (Estimated)
Dates: Start 2022-05-27 (Actual); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-02-01 (Estimated)

PRIMARY OUTCOMES:
Change of e-cigarette use | Baseline
  Measured by the questionnaire including the following items:e-cigarette use, the daily amount of e-cigarette, the age of first e-cigarette use, the reasons for first e-cigarette use, the place where participant first smoked e-cigarette, e-cigarette dependence , the type and amount of other tobacco products used and the daily smoking place.
Change of e-cigarette use | 6 month follow up
  Measured by the questionnaire including the following items:e-cigarette use, the daily amount of e-cigarette, the age of first e-cigarette use, the reasons for first e-cigarette use, the place where participant first smoked e-cigarette, e-cigarette dependence , the type and amount of other tobacco products used and the daily smoking place.
Change of knowledge,attitudes and cognitions related to e-cigarette | Baseline
  The questionnaire items were compiled according to the literature review content, and the questionnaire contained 20 items in total. Six items were related to e-cigarette knowledge, five items are related to the susceptibility of e-cigarettes,eight items are related to the perceived harmfulness of e-cigarettes, one item is related to the perceived relative risk.
Change of knowledge,attitudes and cognitions related to e-cigarette | 6 month follow up
  The questionnaire items were compiled according to the literature review content, and the questionnaire contained 20 items in total. Six items were related to e-cigarette knowledge, five items are related to the susceptibility of e-cigarettes,eight items are related to the perceived harmfulness of e-cigarettes, one item is related to the perceived relative risk.
Change of awareness of new regulations on e-cigarette control | Baseline
  Measured by a yes-or-no question in the questionnaire，and those who answered yes can be considered to be aware of e-cigarette regulations.
Change of awareness of new regulations on e-cigarette control | 6 month follow up
  Measured by a yes-or-no question in the questionnaire，and those who answered yes can be considered to be aware of e-cigarette regulations.

CONTACTS AND LOCATIONS:
Overall Officials: Wei Xia, PhD, Principal Investigator — Sun Yat-sen University
Locations (1):
- XIAW, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
The non-identified individual participant data will be shared after the outcomes have been published.
Supporting Information: SAP
Time Frame: After the publication of the study
Access Criteria: Researchers should contact the PI for approval of the study protocol.